CLINICAL TRIAL: NCT06715956
Title: A Multicenter, Observational Study to Investigate Sputum Inflammation Phenotyping and Predict Clinical Outcomes in Non-Cystic Fibrosis Bronchiectasis, with Subsequent Participation in the HSK31858 Clinical Trial
Brief Title: Observational Study of Sputum Inflammation Phenotypes and Clinical Outcomes in Non-Cystic Fibrosis Bronchiectasis
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Deputy Director of the Clinical Research Center, Guangzhou Institute of Respiratory Disease
Other Study IDs: HSK31858IIT
Record Dates: First submitted 2024-11-24; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Non-cystic Fibrosis Bronchiectasis (NCFBE)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples With DNA — sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Inflammatory Subtype A: Participants classified under this inflammatory subtype based on sputum analysis will be observed without any intervention during the observational phase.
  Interventions: Other: Observational Cohort Classification of Inflammatory Subtypes in Bronchiectasis
- Inflammatory Subtype B: Participants classified under this inflammatory subtype based on sputum analysis will be observed without any intervention during the observational phase.
  Interventions: Other: Observational Cohort Classification of Inflammatory Subtypes in Bronchiectasis
- Inflammatory Subtype C: Participants classified under this inflammatory subtype based on sputum analysis will be observed without any intervention during the observational phase.
  Interventions: Other: Observational Cohort Classification of Inflammatory Subtypes in Bronchiectasis
- Inflammatory Subtype D: Participants classified under this inflammatory subtype based on sputum analysis will be observed without any intervention during the observational phase.
  Interventions: Other: Observational Cohort Classification of Inflammatory Subtypes in Bronchiectasis

INTERVENTIONS:
Other: Observational Cohort Classification of Inflammatory Subtypes in Bronchiectasis — This observational study classifies patients with non-cystic fibrosis bronchiectasis into inflammatory subtypes based on sputum analysis. No active treatment or intervention is administered during this observational phase. Participants will later be considered for treatment with HSK31858 as part of an independent clinical trial.

SUMMARY:
This is an observational, multicenter study aimed at investigating the inflammation phenotypes in sputum samples from patients with non-cystic fibrosis bronchiectasis (NCFBE). The study will observe and classify these phenotypes during the clinical screening phase without any intervention. Patients enrolled in this study may later participate in the HSK31858 clinical trial, where they will receive treatment as part of the trial protocol. After the unblinding of the trial, the study will analyze the relationship between sputum inflammation phenotypes and clinical outcomes, including treatment response and prognosis. The goal is to develop a clinical prediction model that incorporates inflammation subtypes to better predict patient outcomes in bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and BMI≥18.0 kg/m^2 at the time of signing the ICF.
2. Chest HRCT showed bronchiectasis affecting one or more lobes and was confirmed by a clinician as NCFBE(clinically characterized by chronic cough, expectoration and/or intermittent hemoptysis, with or without shortness of breath and respiratory failure). HRCT was considered effective if the patient had received HRCT in the same hospital within 12 months and screening HRCT is not necessary.
3. Have at least 2 pulmonary exacerbations in the past 12 months before Screening.
4. If long-term treatment with bronchodilators (long-acting β-agonists and/or long-acting muscarinic antagonists) is required, the dose and regimen should remain stable for at least 3 months before the screening visit and throughout the study period.
5. The estimated survival time ≥ 12 months.
6. Women must be post-menopausal, surgically sterile, or using highly effective contraception methods from Day 1 to at least 30 days after the last dose.
7. Males with female partners of childbearing potential must be using effective contraception from Day 1 to at least 90 days after the last dose.
8. Give their signed study informed consent to participate.

Exclusion Criteria:

1. Have a primary diagnosis of COPD or asthma as judged by the Investigator. 2. A history of malignancy (excluding cured basal cell carcinoma of the skin, carcinoma in situ, and papillary carcinoma of the thyroid gland. The patients who had survived lung cancer surgery for at least 5 years without antitumor therapy can enroll in the study ) within 5 years prior to screening or a history of antitumor therapy.

3. Have bronchiectasis due to CF (HRCT showed that the above lung diseases became predominant) as judged by the Investigator.

4. Currently being treated Non-tuberculous Mycobacterial (NTM) pulmonary infections, allergic bronchopulmonary aspergillosis, or tuberculosis (TB), or active and currently symptomatic infections caused by COVID-19, or have the history of bronchopulmonary aspergillosis.

5. Patients with severe pulmonary fibrosis such as lung destruction, pneumonectomy surgery history, and pneumoconiosis, as well as previous or existing decompensated stage of pulmonary heart disease.

6. Patients who had experienced any degree of acute exacerbation of bronchiectasis or were developing an acute exacerbation of bronchiectasis before 4 weeks of screening.

7. Patients who had hemoptysis and required medical intervention within 4 weeks prior to screening(except for coughing up minorbloody streaks).

8. Patients previously treated with HSK31858 or other DPP1 inhibitor products. 9. Subjects with uncontrolled hypertension (SBP ≥180 mmHg at rest and/or DBP ≥110 mmHg).

10. Subjects with uncontrolled type 1 or type 2 diabetes (fasting plasma glucose >7.0 mmol/L).

11. Subjects with a history of liver disease or current treatment for liver disease during the screening period, including but not limited to acute or chronic hepatitis, cirrhosis or liver failure (except for mild to moderate non-alcoholic fatty liver disease).

12. Active hepatitis B virus infection (hepatitis B surface antigen positive with HBV-DNA load above the lower limit of detection), active hepatitis C virus infection (HCV antibody positive with HCV-RNA load above the lower limit of detection), or known HIV infection or syphilis infection.

13. Any other unstable clinical condition, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic, psychiatric, or major physiological dysfunction, that the investigator considers to be (a) likely to affect patient safety throughout the study; (b) Influence the results of the study and its interpretation; (c) impeding the patient's ability to complete the entire study.

14. Laboratory tests during the screening period meet the following conditions: AST>2.0×ULN or ALT>2.0×ULN or TBIL>1.5×ULN eGFR<60ml/min/1.73m2 Hb<90 g/L WBC <3×109 /L PLT <70×109 /L INR>1.5ULN，PT>ULN+3s, or APTT>ULN+10s. 15. Had participated in a clinical trial of any other drug or medical device in the 3 months prior to the screening (a drug or medical device treated with a clinical trial) or the subject had not been more than 5 half-lives from the last clinical trial of the drug at the time of screening.

16. Medications that may cause hyperkeratosis (e.g., tumor necrosis factor-α antagonists) within 4 weeks prior to screening.

17. Patients who have used a strong inducer or suppressor of CYP3A within 14 days or 5 half-lives of the first investigational drug (whichever is longer).

18. Patients who had smoked an average of 10 cigarettes or more per day in the previous 1 year were screened.

19. Pregnancy and lactation. 20. The subjects were unable to complete the questionnaires due to their limited educational level, or the subjects and their families failed to fill in the subjects' log cards.

21. Had received live attenuated vaccine within 30 days before randomization. 22. The investigators judged that there were other conditions that were not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 years and older with a confirmed diagnosis of non-cystic fibrosis bronchiectasis (NCFBE).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of pulmonary exacerbations | week 52

SECONDARY OUTCOMES:
Time to first pulmonary exacerbation | week 52
Change from Baseline(Screening) in 24-hour Sputum Weight and Sputum purulence score | week 52
  score from 0 to 8
Change from Baseline in the Respiratory Symptoms Domain Score of the Quality of Life (QOL) Bronchiectasis questionnaire | week 52
  score from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No